CLINICAL TRIAL: NCT02345499
Title: Open Versus Laparoscopic Radical Cystectomy for Invasive Bladder Cancer in the Elderly Patient. A Multicenter Randomized Clinical Trial.
Brief Title: Open Versus Laparoscopic Radical Cystectomy
Acronym: OvsL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Principal Investigator, Pagliarulo Vincenzo, Medical Doctor, Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 4201
Record Dates: First submitted 2015-01-14; First posted 2015-01-26 (Estimated); Last update posted 2015-01-26 (Estimated); Status verified 2015-01

CONDITIONS: Bladder Cancer
Keywords: Radical cystectomy; Laparoscopy
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic radical cystectomy (Experimental): Surgery: Laparoscopic radical cystectomy with open urinary diversion
  Interventions: Procedure: Laparoscopic radical cystectomy with open urinary diversion
- Open radical cystectomy (Active Comparator): Surgery: Open radical cystectomy with open urinary diversion
  Interventions: Procedure: Open radical cystectomy with open urinary diversion

INTERVENTIONS:
Procedure: Laparoscopic radical cystectomy with open urinary diversion — Laparoscopic surgical procedure in which the bladder is removed because of bladder cancer and a urinary diversion is performed
  Arms: Laparoscopic radical cystectomy
Procedure: Open radical cystectomy with open urinary diversion — Open surgical procedure in which the bladder is removed because of bladder cancer and a urinary diversion is performed
  Arms: Open radical cystectomy

SUMMARY:
To date, no trials have been designed to compare open Vs laparoscopic radical cystectomy in the elderly patients, both in terms of functional and clinical outcome measures. A more meaningful comparison of the two modalities is that of a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a histologically proven diagnosis of transitional cell carcinoma of the bladder
2. Patients with an indication to ureterocutaneostomy or ileal conduit
3. ECOG Performance Status ≤ 2
4. WBC count ≥4,000/μL; platelet count ≥150,000/μL

4.Recent (within 6 weeks of cystectomy) total body CT imaging study excluding distant metastases as well as upper urinary tract TCC

Exclusion Criteria:

1. Patients who have previously undergone lower abdominal and/or pelvic surgery for invasive cancer (i.e. radical prostatectomy, large bowel surgeries with or without ileal/colonic conduit)
2. Patients who have previously received any pelvic irradiation
3. Patients with a synchronous upper urinary tract malignancy requiring a nephroureterectomy concomitant to cystectomy
4. Patients candidates for a palliative cystectomy (i.e. recurrent haematuria which cannot be treated by endoscopy)
5. Patients with a histologically proven diagnosis of bladder adenocarcinoma, squamous cell carcinoma, and small cell carcinoma

Min Age: 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2014-01; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Complication rate | 24 months
  Comparison of the complication rate among the two cohorts of patients under investigation according to the Clavien classification.

SECONDARY OUTCOMES:
Health related quality of life | 24 months
  Comparison of health related quality of life among the two cohorts under investigation according to the SF-36 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo VP Pagliarulo, M.D., Principal Investigator — Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari
Locations (1):
- Vincenzo Pagliarulo, Bari, Italy, Italy

REFERENCES:
- [Background] Haber GP, Crouzet S, Gill IS. Laparoscopic and robotic assisted radical cystectomy for bladder cancer: a critical analysis. Eur Urol. 2008 Jul;54(1):54-62. doi: 10.1016/j.eururo.2008.03.076. Epub 2008 Apr 1. PMID 18403100
- [Background] Hemal AK. Robotic and laparoscopic radical cystectomy in the management of bladder cancer. Curr Urol Rep. 2009 Jan;10(1):45-54. doi: 10.1007/s11934-009-0009-8. PMID 19116095
- [Background] Edwards BK, Howe HL, Ries LA, Thun MJ, Rosenberg HM, Yancik R, Wingo PA, Jemal A, Feigal EG. Annual report to the nation on the status of cancer, 1973-1999, featuring implications of age and aging on U.S. cancer burden. Cancer. 2002 May 15;94(10):2766-92. doi: 10.1002/cncr.10593. PMID 12173348
- [Background] Chamie K, Hu B, Devere White RW, Ellison LM. Cystectomy in the elderly: does the survival benefit in younger patients translate to the octogenarians? BJU Int. 2008 Aug;102(3):284-90. doi: 10.1111/j.1464-410X.2008.07636.x. Epub 2008 Apr 11. PMID 18410437
- [Background] Nielsen ME, Shariat SF, Karakiewicz PI, Lotan Y, Rogers CG, Amiel GE, Bastian PJ, Vazina A, Gupta A, Lerner SP, Sagalowsky AI, Schoenberg MP, Palapattu GS; Bladder Cancer Research Consortium (BCRC). Advanced age is associated with poorer bladder cancer-specific survival in patients treated with radical cystectomy. Eur Urol. 2007 Mar;51(3):699-706; discussion 706-8. doi: 10.1016/j.eururo.2006.11.004. Epub 2006 Nov 13. PMID 17113703
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716